CLINICAL TRIAL: NCT06929819
Title: Research on the Safety and Efficacy of Intraoperative Radiation Therapy in Malignant Cerebral Tumor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhang Nu, Discipline Leader of Neurosurgery department, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA [2024]349
Record Dates: First submitted 2024-09-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma; Brain Tumor, Primary; Brain Tumor - Metastatic
Keywords: Brain Tumor; Intraoperative Radiation Therapy
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: This trial is a single-arm study, and patients who are willing to undergo IORT are selected for inclusion in the study after initial screening, and intraoperative radiotherapy of an appropriate dose is given immediately after tumor resection during surgery, followed by postoperative adjuvant therapy according to disease guidelines. The time of recurrence and/or death and the time of adverse events were recorded. This trial is a superiority study and the control is currently the world-recognized median OS or PFS.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Radiation Therapy in Malignant Cerebral Tumor (Experimental)
  Interventions: Radiation: Intraoperative Radiation Therapy in Malignant Cerebral Tumor

INTERVENTIONS:
Radiation: Intraoperative Radiation Therapy in Malignant Cerebral Tumor — This technique can fully expose the tumor bed during the operation, and pull the brain tissue around the tumor under the microscope to de-radiation, so as to exceed the total dose level of standard conformal conventional external radiation therapy (EBRT), maximize the radiobiological effect of a single high-dose irradiation, and deliver precise radiation to the tumor bed, while minimizing the radiation dose of peripheral nerve tissue. This technique is also a good choice for patients with orthotopic recurrent tumors who can no longer tolerate one more EBRT. Intraoperative radiotherapy technology can reduce the chance of postoperative tumor recurrence and improve the survival and prognosis of patients by providing a higher effective total dose to the tumor bed, while promoting dose escalation without significantly increasing the occurrence of complications in normal tissues, and improving the local control rate.

SUMMARY:
According to the latest national cancer statistics released by the National Cancer Center in February 2022, intracranial tumors account for about 60%-70% of the more than 3.5 million cancer patients, and the morbidity and mortality remain high. Intracranial malignant tumors have become a problem that needs to be solved urgently because of their early recurrence, rapid progression, and short survival, and intracranial malignant tumors include high-grade gliomas, metastases, lymphomas, etc.

Glioblastoma (GB) is the most common primary malignancy in the adult central nervous system, accounting for about 57% of all gliomas and 48% of all primary weighted nervous system malignancies. At present, the standard treatment for glioblastoma is mainly surgical treatment, supplemented by postoperative concurrent chemoradiotherapy and adjuvant chemotherapy, but the prognosis of patients is still poor, with a one-year survival rate of 40.6%, a five-year survival rate of only 5.6%, and an average survival time of 12-15 months.

For patients diagnosed with intracranial malignancies (including high-grade glioma, metastases, lymphoma, etc.), multimodal image-guided microsurgery combined with postoperative chemoradiotherapy recommended by the guidelines, and intraoperative radiotherapy with tumor bed radiation therapy to achieve targeted and precise tumor treatment, thereby improving the prognosis of patients (including progression-free survival and median overall survival, etc.)

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, non-pregnant or lactating women
* KPS ≥60
* MRI and CT of the brain with contrast should be considered for diagnosis of high-grade glioma or other malignant brain tumors
* No other underlying diseases that affect survival time, follow-up or quality of life, and no other serious organic lesions
* Not receive radiotherapy, chemotherapy and other treatment methods for intracranial lesions in the past;
* Tumor located supratentorium, and the position should ensure that the tumor resection volume is more than 90%;
* The required dose of standard radiotherapy exceeds normal tissue tolerance
* No related contraindications such as intraoperative radiotherapy and craniotomy.

Exclusion Criteria:

* Refuse to undergo craniotomy or radiation therapy;
* The postoperative paraffin pathological results were not high-grade gliomas or other cranial malignant tumors;
* Refuse to participate in the clinical trial after informed consent without the above exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
The overall survival of enrolled patients was compared with the overall survival reported in the literature | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Nu Zhang, Professor, Principal Investigator — he First Affiliated Hospital of Sun Yat sen University